CLINICAL TRIAL: NCT02362581
Title: Comparison of Prophylaxis and On-demand Treatment in Children With Moderate to Severe Hemophilia A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Darintr Sosothikul, Pediatric Hematology/Oncology department, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3125055
Record Dates: First submitted 2015-01-29; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Prophylaxis; Hemophilia A
Keywords: Prophylaxis treatment; On demand treatment; Severe hemophilia A; Moderate hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- On demand treatment, prophylaxis treatment (Experimental): On demand treatment arm:Patients received factorVIII concentrate(Hemofil M) when they had bleeding episodes.
  Prophylaxis arm: patients received factorVIII concentrate (Hemofil M) 30-35 unit/kg once a week
  Interventions: Other: prophylaxis treatment, on demand treatment

INTERVENTIONS:
Other: prophylaxis treatment, on demand treatment
  Other Names: Hemofil M

SUMMARY:
Comparison of prophylaxis and on-demand treatment in children with moderate to severe hemophilia A.

This study determines to compare the efficacy of prophylaxis and on-demand treatment in moderate to severe hemophilia A children in King Chulalongkorn Memorial Hospital, Bangkok, Thailand

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months to 18 years
* Diagnosis severe and moderate hemophilia A

Exclusion Criteria:

* platelet < 100,000/mm3
* No factor VIII inhibitor

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of bleeding episodes require treatment | one year
number of school days lost | one year
Number of admission days | one year

SECONDARY OUTCOMES:
Joint scores | one year
Quality of life score | one year
Amount of Facter VIII concentration used | one year

CONTACTS AND LOCATIONS:
Overall Officials: Darintr Sosothikul, Asso professer, Principal Investigator — pediatric Hemato-Oncology
Locations (1):
- pediatric Hemato-oncology department, King Chulalongkorn Memorial Hospital, Pratumwan, Bangkok, Thailand